CLINICAL TRIAL: NCT04186975
Title: Computerized Antepartum Monitoring Using Non-invasive Fetal Ecg for High Risk Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Oren Grunwald MD, Oren Grunwald MD, Rambam Health Care Campus
Other Study IDs: 0529-19-RMB
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Cardiotocography
Keywords: FETAL MONITORING, CARDIOTOCOGRAPHY

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-risk pregnant women: Normal cohort: this cohort consists of pregnancies which are not at risk. Data are recorded during the normal checkup happening as part of the usual care pathway
  Interventions: Device: Non-Invasive fetal ECG; Device: Fetal heart rate monitor
- High-risk pregnant women: Risk cohort: this cohort consists of pregnancies at risk and which are regularly recorded for the purpose of fetal surveillance. Specifically, the investigators recruit pregnancies with intra uterine growth restricted fetuses for this study.
  Interventions: Device: Non-Invasive fetal ECG; Device: Fetal heart rate monitor

INTERVENTIONS:
Device: Non-Invasive fetal ECG — Non-Invasive fetal ECG
Device: Fetal heart rate monitor — Fetal heart rate monitor

SUMMARY:
The long term aim of this research is to evaluate a portable NI-FECG (Non-invasive fetal ECG) monitor (Holter NI-FECG) which can be used for regular remote assessment of fetal health in pregnancies at risk or to follow-up on treatments. The elaboration of a NI-FECG Holter device will offer new opportunities for fetal diagnosis and remote monitoring of problematic pregnancies because of its low-cost, non-invasiveness, portability and minimal set-up requirements.

DETAILED DESCRIPTION:
Pregnant patients that are of gestational age in which fetal heart rate monitoring is recommended and feasible will be enrolled to this cohort study. Each patient will be monitored via conventional fetal heart rate monitoring in addition to the NI-FECG method and both methods will be directly compared. Each patient will be her own control. NI-FECG is a non-invasive method of fetal monitoring' thus no ethical issues are relevant. Nevertheless, each patient will sign informed consent before participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies.
* low-risk pregnancy: women from the post-date clinic (after 40 weeks' gestation) in which we perform routinely Non stress test and ultrasound.
* High-risk pregnancy: women who are hospitalized for different indications: IUGR, diabetes, hypertension, non-reassuring fetal heart rate, Decreased fetal movements

Exclusion Criteria:

* Non singleton pregnancies.
* Do not want to participate in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Low risk and High risk pregnancies. Low risk post date patients. High risk intra uterine growth restricted fetuses.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Identification of abnormal fetal heart rate from NI-FECG | 2 years
  To compare the clinical interpretation of the NI-FECG obtained fetal heart rate trace to the fetal heart rate interpretation from the fetal heart rate obtained from conventional CTG. This will involve blinded reading and scoring of FHR obtained from the NI-FECG and CTG from a panel of expert clinician.
Computerized NI-FECG for the prediction of abnormal FHR traces | 2 years
  To compare the computerized analysis of the FHR trace obtained using NI-FECG to the clinician visual interpretation of the FHR trace obtained using CTG (usual care). This will involve the implementation of algorithms that can detect standard14 and new features assessing the Fetal HRV (FHRV) and the elaboration of a machine learning model which can predict abnormal traces from these features
Comparison between computerized CTG and NI-FECG | 4 years
  To compare the predictive power of computerized CTG versus computerized NI-FECG for the assessment of abnormal traces. For that purpose, a machine learning model will be trained (1) on features extracted from the FHR trace obtained using CTG and (2) on features extracted from the FHR obtained using the NI-FECG trace
Develop a portable NI-FECG monitor for remote fetal monitoring. | 4 years
  To develop a portable NI-FECG monitor which can be used to record the fetal ECG at the patient's home. The monitor will transfer the data to a remote server where source separation will be performed to extract the fetal ECG. Algorithms implemented for extracting characteristic features and the machine learning model will be run to predict whether the traces are normal or abnormal. The elaboration of such algorithm is particularly relevant for resource constrained region where medical experts is scarce.

CONTACTS AND LOCATIONS:
Overall Officials: Oren Grunwald, MD, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No